CLINICAL TRIAL: NCT00635947
Title: Randomized Trial of Maternal Hydration on the Increase of Amniotic Fluid Index
Brief Title: Study of Maternal Hydration on the Increase of Amniotic Fluid Index
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Responsible Party: Vera Therezinha Medeiros Borges, Department of Obstetrics and Gynaecology - Botucatu Medical School, UNESP
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-08
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-03-14 (Estimated); Status verified 2008-03

CONDITIONS: Pregnancy
Keywords: Amniotic fluid index; maternal hydration; isotonic solution; Amniotic Fluid
MeSH Terms: interventions — Isotonic Solutions; Water

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): isotonic solution - 1.5L
  Interventions: Other: isotonic solution
- 2 (Active Comparator): water- 1.5L
  Interventions: Other: water
- 3 (Placebo Comparator): water-200mL
  Interventions: Other: water

INTERVENTIONS:
Other: isotonic solution — 1.5 L- during 2-4hours
  Other Names: Isotonic
  Arms: 1
Other: water — 1.5 L- during 2-4hours
  Other Names: Water 1.5
  Arms: 2
Other: water — 200mL- during 2-4hours
  Other Names: Water 200
  Arms: 3

SUMMARY:
The purpose of this study is to determine the effect of maternal hydration with oral isotonic solution and water on amniotic fluid (AF) index in women with normohydramnios.

DETAILED DESCRIPTION:
Objective: To determine the effect of maternal hydration with oral isotonic solution and water on amniotic fluid (AF) index in women with normohydramnios.

Subjects and Methods: Women with normal AF index and gestational age between the 33 and 36 weeks without maternal complications were randomized into three groups (isotonic solution, water, control). The isotonic solution and water groups were instructed to drink 1.5L of respective solution; the control group was instructed to drink 200mL of water. AF index was measured before and after hydration. The investigator performing the AF index was blinded to the subject's group.

Results: Ninety-nine women completed the study without any maternal adverse effects. The mean increase in amniotic fluid index after hydration was significantly greater in the isotonic solution and water groups (12.1mm, p=0.02; 13.1mm, p=0.05; respectively) than the control group (1.4mm, p=0.74). There was no significant difference between the isotonic solution and water groups. Hydration with isotonic solution and water improved the chance of 20% of increase of amniotic fluid index in 10.2 (95% CI 1.9-98.9) and 6.0 (95% CI 1.0-45.5) times respectively.

Conclusion: Maternal hydration with isotonic solution or water increased AF index in women with normohydramnios.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 33 and 36 weeks
* singleton pregnancy
* intact membranes
* initial AF index between 5 and 95 per cent

Exclusion Criteria:

* no maternal complications
* no fetal structural malformation
* no evidence of fetal distress on nonstress test

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 1998-07; Primary Completion 1999-07 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
the effects of maternal oral hydration with isotonic fluid and water on amniotic fluid index in women with normohydramnios | 4horas

SECONDARY OUTCOMES:
compare the effects of maternal oral hydration with isotonic fluid and water on amniotic fluid index in women with normohydramnios | 4horas

CONTACTS AND LOCATIONS:
Overall Officials: Vera M Borges, PhD, Principal Investigator — School of Medicine of Botucatu--São Paulo State University (Unesp)
Locations (1):
- School of Medicine of Botucatu--São Paulo State University (Unesp)--, Botucatu, São Paulo, Brazil

REFERENCES:
- [Result] Kilpatrick SJ, Safford KL, Pomeroy T, Hoedt L, Scheerer L, Laros RK. Maternal hydration increases amniotic fluid index. Obstet Gynecol. 1991 Dec;78(6):1098-102. PMID 1945215
- [Result] Kilpatrick SJ, Safford KL. Maternal hydration increases amniotic fluid index in women with normal amniotic fluid. Obstet Gynecol. 1993 Jan;81(1):49-52. PMID 8416460